CLINICAL TRIAL: NCT01996215
Title: Cognitive Changes and Brain Connectivity in Age-Related Macular Degeneration
Brief Title: Brain Connectivity in Age-Related Macular Degeneration
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Other Study IDs: Pro00046073; R01AG043438 (NIH)
Record Dates: First submitted 2013-11-22; First posted 2013-11-27 (Estimated); Last update posted 2019-02-07 (Actual); Status verified 2018-12

CONDITIONS: Age-Related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- AMD controls
- AMD cases

SUMMARY:
This study is to determine how cognitive deficits (e.g.,verbal fluency deficit) in patients with Age-Related Macular Degeneration (AMD) relate to specific aspects of brain and function. The study team will assess whether the "brain signatures" associated with specific cognitive deficits differ in older adults with and without AMD.

ELIGIBILITY:
Inclusion Criteria:

AMD

- Vision loss attributable to AMD

Controls

* Age match (± 5 yrs)
* Gender match
* Education match (± 4yrs)
* Normal macular exam

Exclusion Criteria:

AMD

* Other significant eye pathology
* Mod/severe dementia
* Communication barrier that precludes testing

Controls

* Other significant eye pathology
* Mod/severe dementia
* Communication barrier that precludes testing

MRI subset

* Devices or material incompatible with 3.0 Tesla MRI
* Conditions that may interfere with interpretation of fMRI (e.g. history of stroke, brain tumor or previous brain surgery; psychoactive medications; seizure disorder)
* Claustrophobia
* Left-handed
* Body weight > 300 lbs
* Pregnant women

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study will include 300 participants: 150 subjects with AMD plus 150 age, gender, and education-matched adults without AMD. All participants will receive baseline and 2 year neurocognitive tests and a subset will provide structural and "resting stage"functional magnetic resonance images (MRIs) at each time point.
Sampling Method: Non-Probability Sample
Enrollment: 238 (Actual)
Dates: Start 2014-04; Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Cognitive Changes and Brain Connectivity in Age-Related Macular Degeneration | Baseline, anticipated 2 years
  All Participants will receive neurocognitive testing, health and lifestyle surveys, audiometry and eye exams. Brain MRIs will be obtained on half the cohort, as this will provide sufficient power to accomplish the Aims that involve neuroimaging data. These MRIs will be obtained while participants are in the "resting state" meaning they are awake but not instructed to perform specific scanner. Two years after baseline exams, participants will return for repeat data collection. Participants who received an MRI at baseline will receive repeat resting-state, brain MRI at 2-year follow-up, unless they have developed contradictions to MRI scans in the interim.

CONTACTS AND LOCATIONS:
Overall Officials: Heather Whitson, MD, Principal Investigator — Duke Medicine
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States